CLINICAL TRIAL: NCT05282992
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate Efficacy and Tolerability of a Food Supplement in Healthy Volunteers With Joint Discomfort
Brief Title: NAtive Collagen Type II In Healthy VoluntEers With Joint Discomfort
Acronym: ACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: PJ-00081
Record Dates: First submitted 2022-02-23; First posted 2022-03-16 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2023-01

CONDITIONS: Joint Pain
MeSH Terms: conditions — Arthralgia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Native type II collagen (Experimental): Native type II collagen
  Interventions: Dietary Supplement: Native type II collagen
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Native type II collagen — 1 capsule/day
  Arms: Native type II collagen
Dietary Supplement: Placebo — 1 capsule/day
  Arms: Placebo

SUMMARY:
Collagen Supplement is a natural ingredient that contains native collagen derived from chicken sternum. Collagen Supplement is efficacious and safe on healthy subjects as compared to placebo.

DETAILED DESCRIPTION:
This study will include 100 healthy volunteers in which will be evaluated if the collagen supplement is able to obtain differences versus placebo in pain and function. It will be a randomized, double-blind, placebo-controlled study with proportion 1:1 between treatments

ELIGIBILITY:
Inclusion Criteria:

* Males and non-pregnant females 30-65 years old with a Body Mass Index (BMI) of approximately 18 to 30 kg/m2. (see Section 4.0)
* Unilateral or bilateral knee discomfort for greater than 3 months.
* VAS score during knee movement between 30-50 mm after 7-day withdrawal of excluded medications.
* Reach joint discomfort of 5/10 on a 11-point Likert scale ( score 0 to 10) within 10 minutes of going up and down stairs.
* Clinical laboratory results that are within normal range or considered not clinically significant by the Principal Investigator.
* Be willing to participate in all scheduled visits, tests, and other trial procedures according to the clinical protocol. To do so and be able of using the fitness tracker, a phone or tablet compatible with the Fitbit app is required. (Apple iOS 12.2 or higher, Android OS 7.0 or higher.)
* Be willing to refrain from taking ibuprofen, aspirin or other Non-steroidal anti-inflammatory drugs (NSAIDs), or any other pain reliever (OTC (Over the Counter) or prescription) during the entire study other than acetaminophen (paracetamol) as rescue medication.
* Provide a signed and dated informed consent indicating that the subject has been informed of all pertinent aspects and possible risks associated with participation in the study.
* Be willing to refrain from taking dietary supplements during the entire study that have any underlying joint benefit (collagen, glucosamine, chondroitin, MSM, Hyaluronic Acid, Turmeric, Natural Eggshell Membrane, Omega-3 fatty acids, PEA, Boswellia,…)

Exclusion Criteria:

* History of hypersensitivity to the rescue medication or any of the products used in the study.
* Requirement of drugs to control joint discomfort.
* Regular drug intake to control any kind of pain.
* History of hypersensitivity to eggs, chicken, or fowl.
* History of Knee OA (OsteoArthritis), inflammatory arthropathy, RA (Rheumatoid Arthritis), OA (VAS score greater than 50), or Systemic Lupus Erythematosus.
* Hyperuricemia (>440 μmol/L), history of gout, or both.
* Exercising (intentionally) for more than 10 hours a week
* High intensity exercise for more than 5 hours a week
* Anticipation of surgery within the next 6 months.
* Recent injury in the target knee (past 4 months).
* History of congestive heart failure.
* Anticipated problems with product consumption.
* Evidence or history of clinically significant haematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, neurologic diseases, or malignancies within the last 5 years.
* High alcohol intake (>2 standard drinks per day) or use of recreational drugs (e.g., cocaine, methamphetamine, marijuana, etc.).
* Females who are pregnant or lactating or planning to become pregnant.
* History of any mental illness that might impair the ability of subjects to provide a written informed consent.
* Use of oral corticosteroid, indomethacin, SYSADOAs (symptomatic slow action drug osteoarthritis) within 3 months of Visit 1; topical treatment with corticosteroids within 1 week of visit 1, and consumption of Omega 3 fatty acids or any other joint health dietary supplements within 2 weeks preceding the treatment period.
* Consumed, ibuprofen, aspirin or other NSAIDS, or any other pain reliever (OTC or prescription), or any natural health product, (excluding vitamins) within 7 days of first visit.
* Consumed acetaminophen (paracetamol) within 48 hours of randomization visit.
* Participation in any clinical trials within 30 days prior to first visit.
* Individuals following an energy restricted diet for weight loss

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-03-03 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2024-03-18 (Actual)

PRIMARY OUTCOMES:
Change in joint discomfort onset | Change in joint discomfort onset at 6 months
  Determine differences from baseline on reaching a joint pain of 5/1 while going up and down stairs (max 10 min).

SECONDARY OUTCOMES:
Joint discomfort | Day 0 to day 60, 90, 120, 180
  Visual Analog Scale (VAS, 0-10cm) pain at rest and during activity. A higher VAS means higher pain levels
Joint function | Day 0 to day 60, 90, 120, 180
  Knee injury and Osteoarthritis Outcome Score (KOOS) test
Time to Joint discomfort | Day 0 to day 60, 90, 120, 180
  Time to joint discomfort and to recover from pain in 3 different exercises
6 minute walking timed test (6MWT) | Day 0 and 180
  Distance a person is capable of walking on a flat, hard surface in 6 minutes
Rescue medication consumption | Day 0 to 180, anytime
  Rescue medication: Paracetamol 500mg. max 2 pills/day
Cartilage turnover biomarkers | Day 0 and 180
  Cartilage turnover biomarkers will be measured in blood and urine (CTX-II, C2C, CPII)

OTHER OUTCOMES:
Daily activity levels | Day 0 to 180, anytime
  A fitness tracker will monitor the steps taken daily
Muscle quality | Day 0 and 180
  Muscle quality will be evaluated by an ultrasound index
Safety assessment | Day 0 to 180, anytime
  Adverse events
Safety assessment | Day 0 to day 60, 90, 120, 180
  Medical exams (weight in kilograms, height in meters, BMI in kg/m^2)
Safety assessment | Day 0 to day 60, 90, 120, 180
  Vital signs (heart rate in bpm and blood pressure mmHg)
Safety assessment | Day 0 and 180
  Laboratory analysis (total blood count, glucose, AST, ALT, Cholesterol, Creatinine, BUN, triglycerides, alkaline phosphatase)

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Poal de Reumatología, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No